CLINICAL TRIAL: NCT01476410
Title: A Phase II Trial of Sequential SGN-35 Therapy With Adriamycin, Vinblastine, and Dacarbazine (S-AVD) for Older Patients With Untreated Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin and Combination Chemotherapy in Treating Older Patients With Previously Untreated Stage II-IV Hodgkin Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northwestern University (Other)
Collaborators: Robert H. Lurie Cancer Center (Other); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 11H01; NCI-2011-00684 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00046908 (Other: Northwestern University IRB)
Record Dates: First submitted 2011-10-18; First posted 2011-11-22 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Adult Lymphocyte Depletion Hodgkin Lymphoma; Adult Lymphocyte Predominant Hodgkin Lymphoma; Adult Mixed Cellularity Hodgkin Lymphoma; Adult Nodular Sclerosis Hodgkin Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage IV Adult Hodgkin Lymphoma
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole; Immunohistochemistry; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (antibody-drug conjugate and combination chemo) (Experimental): LEAD-IN: Patients receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.
  AVD CHEMOTHERAPY: Patients then receive doxorubicin hydrochloride IV, vinblastine IV, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients achieving CR receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: brentuximab vedotin; Drug: doxorubicin hydrochloride; Drug: vinblastine; Drug: dacarbazine; Procedure: quality-of-life assessment; Genetic: DNA analysis; Genetic: RNA analysis; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Other: laboratory biomarker analysis; Other: immunohistochemistry staining method; Genetic: polymorphism analysis

INTERVENTIONS:
Drug: brentuximab vedotin — Given IV
  Other Names: anti-CD30 ADC SGN-35; anti-CD30 antibody-drug conjugate SGN-35; antibody-drug conjugate SGN-35; SGN-35
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: vinblastine — Given IV
  Other Names: Velban; Velsar; VLB
Drug: dacarbazine — Given IV
  Other Names: DIC; DTIC; DTIC-Dome
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Genetic: DNA analysis — Optional correlative studies
Genetic: RNA analysis — Optional correlative studies
Radiation: fludeoxyglucose F 18 — Correlative studies
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Correlative studies
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Other: laboratory biomarker analysis — Optional correlative studies
Other: immunohistochemistry staining method — Optional correlative studies
  Other Names: immunohistochemistry
Genetic: polymorphism analysis — Optional correlative studies

SUMMARY:
This phase II trial studies how well giving brentuximab vedotin together with combination chemotherapy works in treating older patients with previously untreated stage II-IV Hodgkin lymphoma (HL). Monoclonal antibody-drug conjugates, such as brentuximab vedotin, can block cancer growth in different ways by targeting certain cells. Drugs used in chemotherapy, such as doxorubicin hydrochloride, vinblastine, and dacarbazine (AVD), work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving brentuximab vedotin, doxorubicin hydrochloride, vinblastine, and dacarbazine together may kill more cancer cells.

DETAILED DESCRIPTION:
LEAD IN: Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1. Treatment repeats every 21 days for 2 courses in the absence of disease progression or unacceptable toxicity.

AVD CHEMOTHERAPY: Patients then receive doxorubicin hydrochloride IV, vinblastine IV, and dacarbazine IV over 30 minutes on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients achieving CR receive brentuximab vedotin IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care
* Previously untreated classical Hodgkin lymphoma (i.e., nodular sclerosis, mixed cellularity, lymphocyte depleted, lymphocyte-rich, and not otherwise specified [NOS]); nodular lymphocyte predominant Hodgkin lymphoma is not eligible
* Stage II, III, and IV disease by Ann Arbor classification
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2
* Patients must have bi-dimensional measurable disease documented in the lymphoma baseline tumor assessment form within 30 days prior to registration (at least 1.5 cm); patients with non-measurable disease in addition to measurable disease must have been assessed within 60 days prior to registration
* Patients must have a bone marrow biopsy (bilateral preferred, unilateral acceptable) within 60 days prior to registration
* Patients must have a multi gated acquisition scan (MUGA) or echocardiogram within 60 days prior to study registration and the ejection fraction must be >= 45%
* Absolute neutrophil count (ANC) > 1000/mm^3
* Platelet count > 75,000/mm^3
* Creatinine < 2.5 mg/dl
* Bilirubin < 3.0 mg/dl
* Patients with documented marrow involvement by lymphoma at the time of registration are not required to meet the above hematologic parameters
* Patients must not have received prior chemotherapy or radiation therapy for the treatment of Hodgkin lymphoma
* Both females and males who have partners of childbearing potential must agree to use an effective contraceptive method during the study and for 30 days following the last dose of study drug
* Patients must sign the informed consent form before registration

Exclusion Criteria:

* Previous treatment with brentuximab vedotin or any other prior anti-CD30-based antibody therapy
* History of another primary malignancy that has not been in remission for at least 3 years; (the following are exempt from the 3-year limit: early stage [stage I or II] breast cancer treated with surgery and radiation +/- hormones [without adjuvant chemotherapy], non-melanoma skin cancer, fully excised melanoma in situ [stage 0], curatively treated localized prostate cancer, and cervical carcinoma in situ on biopsy or a squamous intraepithelial lesion on Papanicolaou test [PAP smear])
* Known cerebral/meningeal disease
* Any active systemic viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy within 1 week prior to first dose
* Patients with hepatitis B surface antigen (HBsAg) positive hepatitis B virus (HBV) infection; patients with prior history of hepatitis B infection, but immune, with only Immunoglobulin G (IgG) hepatitis core antibody + (HBcAb +) must receive anti-viral prophylaxis (e.g., lamivudine 100mg orally [po] daily) for at least 1 week prior to cycle 1 and throughout induction and continuation therapy and for at least 6 months after the last brentuximab vedotin dose; in addition, consultation with a hepatologist is recommended
* Patients with a known hypersensitivity to any excipient contained in the drug formulation
* Patients with dementia or an altered mental state that would preclude the understanding and rendering of informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Overall response rate after chemotherapy | 2 years
  The primary objective of this study is to assess the overall response rate among older patients with HL receiving sequential brentuximab vedotin therapy with AVD chemotherapy

SECONDARY OUTCOMES:
Overall response rate | Baseline, every 3 weeks during the first 2 cycles, every 2 weeks during next 6 cycles, every 4 weeks furing the last 4 cycles, and then every 3 months for up to 3 years from entering the study
  Overall response rate progression-free survival (PFS), time to treatment failure (TTF), freedom from progression (FFP), and overall survival (OS) rates following SGN-35/AVD sequential therapy.
Overall response rate based on best response (CR and PR) and the tumor local control rate (CR, PR, and stable disease [SD]) | Baseline, every 3 weeks during the first 2 cycles, every 2 weeks during next 6 cycles, every 4 weeks furing the last 4 cycles, and then every 3 months for up to 3 years from entering the study
  Estimates of response rate based on best response (CR and PR) and the tumor local control rate (CR, PR, and stable disease [SD])

CONTACTS AND LOCATIONS:
Overall Officials: Leo Gordon, MD, Principal Investigator — Northwestern University
Locations (7):
- United States (7):
  - Stanford University Medical Center, Stanford, California
  - NorthwesternU, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Tufts Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan- Kettering Cancer Center, New York, New York
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Evens AM, Advani RH, Helenowski IB, Fanale M, Smith SM, Jovanovic BD, Bociek GR, Klein AK, Winter JN, Gordon LI, Hamlin PA. Multicenter Phase II Study of Sequential Brentuximab Vedotin and Doxorubicin, Vinblastine, and Dacarbazine Chemotherapy for Older Patients With Untreated Classical Hodgkin Lymphoma. J Clin Oncol. 2018 Oct 20;36(30):3015-3022. doi: 10.1200/JCO.2018.79.0139. Epub 2018 Sep 4. PMID 30179569